CLINICAL TRIAL: NCT01998841
Title: A Double-Blind, Placebo-Controlled Parallel-Group Study in Preclinical PSEN1 E280A Mutation Carriers Randomized to Crenezumab or Placebo, and in Non-Randomized, Placebo-Treated Non-Carriers From the Same Kindred, to Evaluate the Efficacy and Safety of Crenezumab in the Treatment of Autosomal-Dominant Alzheimer's Disease
Brief Title: A Study of Crenezumab Versus Placebo in Preclinical Presenilin1 (PSEN1) E280A Mutation Carriers to Evaluate Efficacy and Safety in the Treatment of Autosomal-Dominant Alzheimer's Disease (AD), Including a Placebo-Treated Non-Carrier Cohort
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Banner Alzheimer's Institute (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN28352
Record Dates: First submitted 2013-11-22; First posted 2013-12-02 (Estimated); Results first posted 2023-09-22 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — crenezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mutation Carriers: Crenezumab (Experimental): Study Period A: Participants will receive Crenezumab subcutaneously (every 2 weeks) or intravenously (every 4 weeks) for at least 260 weeks.
  Study Period B: Participants will be offered the opportunity to continue to receive blinded study drug until the results of the study are known and post-trial access to Crenezumab is started or development of Crenezumab is discontinued.
  Interventions: Drug: Crenezumab
- Mutation Carriers: Placebo (Placebo Comparator): Study Period A: Participants will receive Placebo subcutaneously (every 2 weeks) or intravenously (every 4 weeks) for at least 260 weeks.
  Study Period B: All mutation carriers entering Study Period B will, receive Crenezumab until the results of the study are known and post-trial access to Crenezumab is started or development of Crenezumab is discontinued.
  Interventions: Drug: Placebo
- Non-carriers of Mutation: Placebo (Placebo Comparator): Study Period A: Participants will receive Placebo subcutaneously (every 2 weeks) or intravenously (every 4 weeks) for at least 260 weeks.
  Study Period B: All non-mutation carriers entering Study Period B will continue to receive Placebo, until the results of the study are known and post trial access to Crenezumab is started or development of Crenezumab is discontinued.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Crenezumab — Crenezumab will be administered as per the schedule specified in the treatment arm.
  Other Names: MABT5102A
  Arms: Mutation Carriers: Crenezumab
Drug: Placebo — Placebo will be administered as per the schedule specified in the treatment arm.
  Arms: Mutation Carriers: Placebo; Non-carriers of Mutation: Placebo

SUMMARY:
This study consists of 2 periods: [1] Study Period A - evaluating the efficacy and safety of Crenezumab versus Placebo in participants who carry the PSEN1 E280A autosomal-dominant mutation and do not meet the criteria for mild cognitive impairment due to AD or dementia due to AD and are thus, in a preclinical phase of AD. Participants will be randomised in a 1:1 ratio to receive either Crenezumab or Placebo subcutaneously (every 2 weeks) or intravenously (every 4 weeks) for at least 260 weeks. A cohort of participants (non-mutation carriers) will also be enrolled and will be dosed solely on Placebo and [2] Study Period B - Participants will be offered the opportunity to continue to receive study drug until the results of the study are known and post trial access to Crenezumab is started or development of Crenezumab is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Membership in PSEN1 E280A mutation carrier kindred
* Agrees to conditions of, and is willing to undergo, genetic testing (for example [e.g.], apolipoprotein E [APOE], PSEN1 E280A, and other genetic testing)
* PSEN1 E280A mutation carrier or non-carrier status has been confirmed prior to or during the screening period
* Mini-Mental Stage Examination (MMSE) greater than or equal to (>=) 24 for participants with less than (<) 9 years of education or MMSE >=26 for participants with 9 or more years of education
* Does not meet criteria for dementia due to AD per the National Institute on Aging and the Alzheimer's Association Workgroup (McKhann et al. 2011) criteria
* Does not meet criteria for mild cognitive impairment (MCI) due to AD per the National Institute on Aging and the Alzheimer's Association Workgroup (Albert et al. 2011) criteria
* Adequate vision and hearing in the investigator's judgment to be able to complete testing
* If female, and not documented (by medical records or physician's note) to be surgically sterile (absence of ovaries and/or uterus) or postmenopausal, willing to undergo pregnancy tests at protocol-specific timepoints
* For women who are not documented (by medical records or physician's note) to be surgically sterile (absence of ovaries and/or uterus) or postmenopausal, agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of <1 percent (%) per year (e.g., hormonal implants, combined oral contraceptives, vasectomized partner, tubal ligation) during the treatment period and for at least 16 weeks after the last dose of study drug
* For men with partners of childbearing potential (that is [i.e.], women who are not surgically sterile and are not postmenopausal), agreement to remain abstinent or use a condom as a method of contraception during the treatment period and for at least 8 weeks after the last dose of study drug
* Study partner who agrees to participate in the study and is capable of and willing to: accompany the participant to all required visits; provide information for required telephone assessments; spend sufficient time with the participant to be familiar with his/her overall function and behavior and be able to provide adequate information about the participant including knowledge about domestic activities, hobbies, routines, social skills and basic activities of daily life; work and educational history; cognitive performance including memory abilities, language abilities, temporal and spatial orientation, judgment and problem solving; emotional and psychological state; and general health status
* Participant and study partner have evidence of adequate premorbid functioning (e.g., intellectual, visual, and auditory) and are fluent in, and able to read, the language in which study assessments are administered
* Willing and able to undergo neuroimaging (PET and MRI)
* Serum thyroid stimulating hormone (TSH) and B12 levels within normal or expected ranges for the testing laboratory or if TSH and B12 values are out of range they are judged by the investigator not to be clinically significant. If participant is undergoing thyroid replacement therapy, TSH levels must be within normal or expected ranges for the testing laboratory or, if TSH values are out of range, they do not require any therapeutic actions (treatment or surveillance). If participant is receiving vitamin B12 injections or oral vitamin B12 therapy, B12 levels must be at or above the lower limit of normal for the testing laboratory or, if B12 values are out of range, they do not require any therapeutic actions (treatment or surveillance)
* In good general health with no known co-morbidities expected to interfere with participation in the study

Exclusion Criteria:

* Significant medical, psychiatric, or neurological condition or disorder documented by history, physical, neurological, laboratory, or electrocardiogram (ECG) examination that would place the participant at undue risk in the investigator's judgment or impact the interpretation of efficacy
* History of stroke. Participants with a history of transient ischemic attack may be enrolled if the event occurred >=2 years prior to screening
* History of severe, clinically significant (persistent neurological deficit or structural brain damage) central nervous system trauma (e.g. cerebral contusion)
* Body weight <45 or >120 kilograms (kg)
* History or presence of atrial fibrillation that poses a risk for future stroke in the investigator's judgment
* Clinically significant laboratory or ECG abnormalities (e.g., abnormally prolonged or shortened QTc interval) in the investigator's judgment
* Current presence of bipolar disorder or other clinically significant major psychiatric disorder according to Diagnostic and Statistical Manual of Mental Disorders 4th Edition Text Revision (DSM-IV-TR) or symptom (e.g., hallucinations, agitation, paranoia) that could affect the participant's ability to complete evaluations
* Clinically significant depression, based in part by a Geriatric Depression Scale (short form) (15-point scale) score >9 at screening
* History of seizures (excluding febrile seizures of childhood, or other isolated seizure episodes that were not due to epilepsy in the judgment of the investigator, and required at most time-limited anticonvulsant treatment, and which occurred more than 7 years prior to the screening visit)
* Myocardial infarction within 2 years, congestive heart failure, atrial fibrillation, or uncontrolled hypertension
* Pregnant or nursing women, or women who intend to become pregnant or to nurse infants during the conduct of this trial
* Clinically significant infection within the last 30 days prior to screening
* Positive urine test for drugs of abuse at screening
* History of alcohol or substance dependence within the previous two years
* Use of any other medications with the potential to significantly affect cognition; intermittent or short-term use of these medications may be allowed if deemed medically necessary for the treatment of a non-excluded medical condition with approval from the Medical Monitor. In addition, use of tricyclic antidepressants or benzodiazepines will be permitted if used in stable, low doses for the treatment of a non-excluded medical condition with approval from the Medical Monitor
* Use of typical anti-psychotics or barbiturates
* Use of non-anti-cholinergic antidepressant medications or atypical anti-psychotics unless maintained on a stable dose regimen for at least 6 weeks prior to screening
* Use of any Food and Drug Administration (FDA)/Instituto Nacional de Vigilancia de Medicamentos y Alimentos (INVIMA)-approved medications for treatment of late onset Alzheimer's disease (LOAD) at screening/baseline. Cholinesterase inhibitors and/or memantine are prohibited during the study except in participants enrolled in the study that develop AD dementia
* Use of anti-coagulant medication (heparinoids, heparin, warfarin, thrombin inhibitors, Factor Xa inhibitors), or known coagulopathy or platelet count <100,000 cells/microliter, within 4 weeks of the screening visit; Anti-platelet medications (e.g., aspirin, clopidigrel, dipyridamole) are permitted if on a stable dose for 4 or more weeks prior to screening. Short-term, peri-operative use of anti-coagulants may not result in discontinuation from the study; however, any such use must be discussed with the Medical Monitor
* Treatment with any biologic therapy within five half-lives or 3 months prior to screening, whichever is longer, with the exception of routinely recommended vaccinations, which are allowed
* Use of anti-seizure medication (except in childhood for febrile seizures or if used for non-seizure indications), anti-parkinsonian, or stimulant (e.g., methylphenidate) medications
* Use of investigational drug, device, or experimental medication within 60 days (or five half-lives, whichever is longer) of the screening visit
* Previous treatment with crenezumab or any other therapeutic that targets A-beta
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins
* Contraindication to MRI scan procedures or clinically significant claustrophobia that would contraindicate a brain MRI scan
* Contraindication to PET scan procedures

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Colombia (4):
  - Fundacion Cardiomet, Armenia
  - Clínica de Marly, Bogotá
  - Grupo Neurociencias de Antioquia, Medellín
  - Hospital San Juan de Dios, Yarumal

REFERENCES:
- [Derived] Tariot PN, Lopera FS, Rios-Romenets S, Sink KM, Giraldo-Chica M, Acosta-Baena N, Villegas G, Espinosa A, Castano ML, Munoz C, Ospina P, Bocanegra Y, Tirado V, Henao E, Cardona E, Luna E, Lopez H, Sanchez G, Collazos MM, Alvarez S, Aguillon D, Hu N, Clayton D, Bittner T, Schneider A, Dolton M, Poon V, Nguyen J, Thomas RG, Schneider LS, Chen K, Su Y, Alexander RC, Quiroz YT, Cai Y, Xu YR, Ostaszewski B, Selkoe DJ, Ashton NJ, Denkinger MN, Jakimovich LJ, Doody RS, Langbaum JB, Reiman EM. Safety and efficacy of crenezumab in cognitively unimpaired carriers of the PSEN1Glu280Ala mutation at risk for autosomal-dominant Alzheimer's disease in Colombia (API ADAD Colombia Trial): a phase 2, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2026 Feb;25(2):147-159. doi: 10.1016/S1474-4422(25)00426-0. PMID 41579901
- [Derived] Ghisays V, Lopera F, Goradia DD, Protas HD, Malek-Ahmadi MH, Chen Y, Devadas V, Luo J, Lee W, Baena A, Bocanegra Y, Guzman-Velez E, Pardilla-Delgado E, Vila-Castelar C, Fox-Fuller JT, Hu N, Clayton D, Thomas RG, Alvarez S, Espinosa A, Acosta-Baena N, Giraldo MM, Rios-Romenets S, Langbaum JB, Chen K, Su Y, Tariot PN, Quiroz YT, Reiman EM; API ADAD Colombia Trial Group. PET evidence of preclinical cerebellar amyloid plaque deposition in autosomal dominant Alzheimer's disease-causing Presenilin-1 E280A mutation carriers. Neuroimage Clin. 2021;31:102749. doi: 10.1016/j.nicl.2021.102749. Epub 2021 Jul 4. PMID 34252876
- [Derived] Ramirez Aguilar L, Acosta-Uribe J, Giraldo MM, Moreno S, Baena A, Alzate D, Cuastumal R, Aguillon D, Madrigal L, Saldarriaga A, Navarro A, Garcia GP, Aguirre-Acevedo DC, Geier EG, Cochran JN, Quiroz YT, Myers RM, Yokoyama JS, Kosik KS, Lopera F. Genetic origin of a large family with a novel PSEN1 mutation (Ile416Thr). Alzheimers Dement. 2019 May;15(5):709-719. doi: 10.1016/j.jalz.2018.12.010. Epub 2019 Feb 10. PMID 30745123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were carriers and non-carriers of presenilin 1 (PSEN1) E280A mutation of autosomal-dominant Alzheimer's disease (ADAD) took part in the study at four investigative sites in Colombia from 20 December 2013 to 08 August 2023.
Pre-assignment Details: 252 participants were enrolled to receive their assigned treatment. Study consisted of 2 periods: Study Period A & B. Participants who completed Study Period A had an option to continue treatment in Study Period B. 74 participants from Crenezumab - Mutation Carriers arm, 73 from Placebo - Mutation Carrier arm, and 72 from Placebo - Non-Carriers of Mutation arm choose to continue treatment in Period B.
Groups:
- Study Period A: Crenezumab - Mutation Carriers: Participants who were PSEN1 E280A mutation carriers, received crenezumab, 720 milligrams (mg), subcutaneously (SC), every two weeks (Q2W), or 60 milligrams per kilograms (mg/kg), intravenously (IV), every four weeks (Q4W), for a minimum of 260 weeks during Period A.
- Study Period A: Placebo - Mutation Carrier: Participants who were PSEN1 E280A mutation carriers, received crenezumab matching placebo SC, Q2W, or IV, Q4W, for a minimum of 260 weeks during Period A.
- Study Period A: Placebo - Non-Carriers of Mutation: Participants who were non-carriers of PSEN1 E280A mutation, received crenezumab matching placebo, SC, Q2W or IV, Q4W for a minimum of 260 weeks during Period A.
- Study Period B: Crenezumab: Participants who were PSEN1 E280A mutation carriers and who completed treatment with crenezumab or placebo in Period A were given an option to continue receiving crenezumab, 720 mg, SC, Q2W, or 60 mg/kg, IV, Q4W in Period B for up to 51 weeks.
- Study Period B: Placebo: Participants who were non-carriers of PSEN1 E280A mutation and who received crenezumab matching placebo in Period A were given the option to continue receiving crenezumab matching placebo SC, Q2W or IV, Q4W in Study Period B, for up to 51 weeks.
Period: Study Period A
Arm/Group | Study Period A: Crenezumab - Mutation Carriers | Study Period A: Placebo - Mutation Carrier | Study Period A: Placebo - Non-Carriers of Mutation | Study Period B: Crenezumab | Study Period B: Placebo
Started | 85 | 84 | 83 | 0 | 0
Completed | 79 | 78 | 80 | 0 | 0
Not Completed | 6 | 6 | 3 | 0 | 0
Not completed — Reason Not Disclosed to Prevent Genetic Unblinding | 6 | 6 | 3 | 0 | 0
Period: Study Period B
Arm/Group | Study Period A: Crenezumab - Mutation Carriers | Study Period A: Placebo - Mutation Carrier | Study Period A: Placebo - Non-Carriers of Mutation | Study Period B: Crenezumab | Study Period B: Placebo
Started | 0 (Following the end of Period A participants were given the option to continue receiving treatment in Period B.) | 0 (Following the end of Period A participants were given the option to continue receiving treatment in Period B.) | 0 (Following the end of Period A participants were given the option to continue receiving treatment in Period B.) | 147 (A total of 147 mutation carriers choose to continue receiving treatment in Period B.) | 72 (A total of 72 non-carriers of mutation choose to continue receiving treatment in Period B.)
Completed | 0 | 0 | 0 | 140 | 70
Not Completed | 0 | 0 | 0 | 7 | 2
Not completed — Reason Not Disclosed to Prevent Genetic Unblinding | 0 | 0 | 0 | 7 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants whether or not the participants received the assigned study treatment.
Groups:
- Study Period A: Crenezumab - Mutation Carrier: Participants who were PSEN1 E280A mutation carriers, received crenezumab, 720 mg, SC, Q2W, or 60 mg/kg, IV, Q4W, for a minimum of 260 weeks during Period A.
- Study Period A: Placebo - Mutation Carriers: Participants who were PSEN1 E280A mutation carriers, received crenezumab matching placebo, SC, Q2W or IV, Q4W for a minimum of 260 weeks during Period A.
- Total: Total of all reporting groups
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers | Study Period A: Placebo - Non-Carriers of Mutation | Total
Number analyzed (Participants) | 85 | 84 | 83 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (5.3) | 36.9 (6.3) | 43.3 (7.2) | 39.0 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 59 | 57 | 160
  Male | 41 | 25 | 26 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 85 | 84 | 83 | 252
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 3 | 6 | 15
  Black or African American | 4 | 1 | 1 | 6
  White | 37 | 40 | 35 | 112
  More than one race | 25 | 24 | 33 | 82
  Others | 13 | 16 | 8 | 37

OUTCOME MEASURES:

1. Primary Outcome: Period A: Annualized Rate of Change in the Autosomal-Dominant Alzheimer's Disease (API ADAD) Composite Cognitive Test Total Score
Description: API ADAD Composite Cognitive Test is a combination of tests, most sensitive to detect cognitive decline & progression. API ADAD Composite Cognitive Test total score were computed from: Consortium to Establish a Registry for AD (CERAD) Word List: Recall (score range=0-10); Multilingual Naming Test (score range=0-15); Mini-Mental State Examination (MMSE) for orientation to time (score range=0-5); CERAD Constructional Praxis (measure of visuospatial ability) (score range=0-11); Raven's Progressive Matrices (measure of nonverbal fluid reasoning & visuospatial abilities), Set A (score range=0-12). ADAD-API Cognitive Composite Test total score = [(Multilingual Naming Test Score/15)+(MMSE Score/5)+(Raven's Progressive Matrices Score/12)+(CERAD Word List Recall Score/10)+(CERAD Constructional Praxis Score/11)]*20. Total score ranges=0-100. Higher score=better results. Annualized rate of change in API ADAD Composite Cognitive Test was estimated using random coefficient regression model.
Time Frame: Baseline up to approximately Week 416
Population: Modified Intent-to-Treat (mITT) population included all randomized participants who were mutation carriers and were treated with any amount of study drug.
Measure: Mean (Standard Error); unit: points on scale per year
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers
Number analyzed (Participants) | 84 | 84
points on scale per year | -1.10 (0.29) | -1.42 (0.29)
Statistical Analysis 1: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Analysis was based on random coefficient regression model (RCRM) using unstructured covariance matrix: API Composite Endpoint=Treatment * Analysis Year + interactive voice or Web-based response system (IxRS) defined Age Group + IxRS defined Education History + IxRS defined apolipoprotein E4 (APOE4) Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p = 0.43, RCRM; Difference in Annualized Rate of Change = 0.33, 95% CI 2-sided [-0.48 to 1.13], Standard Error of Mean 0.41

2. Primary Outcome: Period A: Annualized Rate of Change in an Episodic Memory Measure: Free and Cued Selective Reminding Task (FCSRT) Cueing Index
Description: FCSRT assesses immediate & delayed verbal episodic memory, using Controlled Learning to optimize encoding specificity for more effective recall. Participants were to remember a list of 16 items presented on cards. Participant's task was to learn & attempt a free recall of the items, followed by a semantically cued recall of items not spontaneously produced during free recall. There were a total of three learning trials, each preceded by 20 seconds of interfering cognitive task. For first two trials, participants were reminded of any item not recalled in cued recall. Free recall (score range: 0-48) & cued recall (score range: 0-64) assessment occurred immediately, after each of three learning trials, & after a delay of approx. 30 minutes. Higher scores indicate better performance. FCSRT Cueing Index=(FCSRT Total Free Recall score-FCSRT Total Recall score)/(FCSRT Total Free Recall score-48). Score range for FCSRT Cueing Index is 0-1, with higher score=better results.
Time Frame: Baseline up to approximately Week 416
Population: mITT population included all randomized participants who were mutation carriers and were treated with any amount of study drug.
Measure: Mean (Standard Error); unit: points on scale per year
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers
Number analyzed (Participants) | 84 | 84
points on scale per year | -0.03 (0.004) | -0.04 (0.004)
Statistical Analysis 1: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Analysis was based on RCRM using unstructured covariance matrix: FCSRT Cueing Index = Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p = 0.16, RCRM; Difference in Annualized Rate of Change = 0.008, 95% CI 2-sided [-0.003 to 0.02], Standard Error of Mean 0.006

3. Secondary Outcome: Period A: Time to Progression From Preclinical AD to Mild Cognitive Impairment (MCI) Due to AD or From Preclinical AD to Dementia Due to AD
Description: Time to progression was calculated from the time at baseline to first confirmed diagnosis of progression from preclinical AD to MCI or from preclinical AD to dementia due to AD whichever occurred first. Preclinical AD was defined as participants who were at certain risk of developing AD dementia but did not have overt symptoms and did not meet criteria for MCI or dementia.
Time Frame: Baseline up to approximately Week 416
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers
Number analyzed (Participants) | 84 | 84
days | NA [NA to NA] — Median, upper and lower limit of 95% confidence interval (CI) were not estimable due to insufficient number of participants with events. | NA [2622.0 to NA] — Median and upper limit of 95% CI were not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Stratification factors used: Age Group, Education History, APOE4 Carrier Status, Clinical Dementia Rating (CDR) Global Score; Test type: Superiority; p = 0.48, Stratified Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.41 to 1.52] — Hazard ratios were estimated by Cox regression

4. Secondary Outcome: Period A: Time to Progression to Non-zero in CDR Scale Global Score
Description: Time to progression was defined as the time at baseline to first increase in the CDR global score i.e., score of > zero on the CDR Global scale. The standard CDR global scale describes five degrees of impairment in performance on each of six categories of cognitive functioning, including memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. The ratings of degree of impairment obtained on each of the six categories of function was synthesized into one global rating of dementia with a score ranging from 0 to 3 (0 = no dementia, 0.5 = questionable dementia, 1 = mild dementia, 2 = moderate dementia, 3 = severe dementia). A higher score indicates a greater degree of impairment.
Time Frame: Baseline up to approximately Week 416
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers
Number analyzed (Participants) | 84 | 84
days | 2759.0 [2391.0 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [2395.0 to NA] — Median and upper limit of 95% CI were not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Stratification factors used: Age Group, Education History, APOE4 Carrier Status; Test type: Superiority; p = 0.76, Stratified Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.53 to 1.59] — Hazard ratios were estimated by Cox regression

5. Secondary Outcome: Period A: Annualized Rate of Change in the CDR Scale - Sum of Boxes (SOB)
Description: The CDR-SB is a rater administered scale and impairment is scored in the following categories: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care. Impairment was scored on a scale in which no dementia = 0, questionable dementia = 0.5, mild dementia = 1, moderate dementia = 2 and severe dementia = 3. The 6 individual category ratings, or "box scores", were added together to give the CDR-Sum of Boxes which ranges from 0-18, with higher scores indicating greater impairment. Annualized rate of change in CDR Scale - SOB was calculated using RCRM.
Time Frame: Baseline up to approximately Week 416
Population: as for outcome 2
Measure: Mean (Standard Error); unit: points on scale per year
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers
Number analyzed (Participants) | 84 | 84
points on scale per year | 0.30 (0.06) | 0.33 (0.06)
Statistical Analysis 1: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Analysis was based on RCRM using unstructured covariance matrix: CDR-SB = Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p = 0.64, RCRM; Difference in Annualized Rate of Change = -0.03, 95% CI 2-sided [-0.15 to 0.09], Standard Error of Mean 0.06

6. Secondary Outcome: Period A: Annualized Rate of Change in a Measure of Overall Neurocognitive Functioning: RBANS
Description: RBANS is a clinical tool designed to detect and characterize the earliest neurocognitive changes associated with dementia. The RBANS comprised of 12 subtests which generates age-adjusted index scores for five neurocognitive domains: Immediate Memory, Visuospatial/Constructional, Language, Attention and Delayed Memory, which are used to calculate a Total Scale Index score. RBANS Total Score = Index Score based on the (Index Score for Immediate Memory + Index Score for Visuospatial/Constructional + Index Score for Language + Index Score for Attention + Index Score for Delayed Memory). Index scores and total scores range from 40-160. A higher score indicates better cognitive functioning. Annualized rate of change in RBANS was calculated using RCRM.
Time Frame: Baseline up to approximately Week 416
Population: as for outcome 2
Measure: Mean (Standard Error); unit: points on scale per year
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers
Number analyzed (Participants) | 84 | 84
points on scale per year | -0.23 (0.21) | -0.40 (0.21)
Statistical Analysis 1: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Analysis was based on RCRM using unstructured covariance matrix: RBANS Total Score = Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p = 0.55, RCRM; Difference in Annualized Rate of Change = 0.18, 95% CI 2-sided [-0.40 to 0.75], Standard Error of Mean 0.29

7. Secondary Outcome: Period A: Annualized Rate of Change in Mean Cerebral Fibrillar Amyloid Accumulation Using Florbetapir Positron Emission Tomography (PET)
Description: Amyloid deposition in brain is one of the defining neuropathologic findings of AD. Cerebral amyloid burden & effect of crenezumab on cerebral amyloid were assessed using 18F- Florbetapir PET. Florbetapir exhibits high affinity specific binding to amyloid plaques, which allows for a measurement of the relative amyloid burden as the ratio of the standard uptake values (SUVR) in a cortical composite region of interest (including the frontal, temporal, parietal, and cingulate cortices with a subcortical white matter reference region). Annualized rate of change in cerebral fibrillar amyloid accumulation was calculated using RCRM.
Time Frame: Baseline up to approximately Week 416
Population: as for outcome 2
Measure: Mean (Standard Error); unit: SUVR per year
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers
Number analyzed (Participants) | 84 | 84
SUVR per year | 0.017 (0.001) | 0.017 (0.001)
Statistical Analysis 1: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Analysis was based on RCRM using unstructured covariance matrix: PET SUVR = Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p = 0.69, RCRM; Difference in Annualized Rate of Change = -0.0006, 95% CI 2-sided [-0.0037 to 0.0024], Standard Error of Mean 0.002

8. Secondary Outcome: Period A: Annualized Rate of Change in Regional Cerebral Metabolic Rate of Glucose (CMRgI) Using Fluorine-18-Labeled 2-Deoxyglucose (FDG)-PET in a Predefined ROI
Description: Regional CMRgl and the effect of crenezumab on regional CMRgl was assessed using FDG-PET. FDG PET evaluates the regional brain metabolic rates for glucose as a sensitive, in vivo metabolic index of brain function. Regional CMRgl was derived from FDG PET images using an empirically predefined statistical ROI (sROI) known to be preferentially affected by CMRgl decline in participants with AD. Results are reported as standardized uptake value ratios. Annualized rate of change in CMRgI was calculated using RCRM.
Time Frame: Baseline up to approximately Week 416
Population: as for outcome 2
Measure: Mean (Standard Error); unit: SUVR per year
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers
Number analyzed (Participants) | 84 | 84
SUVR per year | -0.012 (0.002) | -0.015 (0.002)
Statistical Analysis 1: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Analysis was based on RCRM using unstructured covariance matrix: FDG-PET = Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p = 0.25, RCRM; Difference in Annualized Rate of Change = 0.003, 95% CI 2-sided [-0.002 to 0.007], Standard Error of Mean 0.002

9. Secondary Outcome: Period A: Annualized Rate of Change in Brain Atrophy Measured by Volumetric Measurements Using Magnetic Resonance Imaging (MRI)
Description: Cerebral atrophy correlates closely with the gradual cognitive decline in AD and can be visualized by MRI. The change in brain atrophy after treatment with crenezumab was measured by volumetric measurements using MRI which measures volumes of the key brain structures-hippocampus, ventricles, and other brain structures-and compares the volumes to standard norms based on the age, gender and cranial volume. The regions of interest for atrophy measurement included whole brain, bilateral hippocampus, and bilateral ventricles. The annualized rate of change in brain atrophy was calculated using RCRM.
Time Frame: Baseline up to approximately Week 416
Population: as for outcome 2
Measure: Mean (Standard Error); unit: cubic millimeter (mm^3)/year
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers
Number analyzed (Participants) | 84 | 84
cubic millimeter (mm^3)/year
  Whole Brain | -721.91 (65.33) | -829.69 (65.42)
  Bilateral Hippocampus | -92.62 (12.25) | -102.22 (12.27)
  Bilateral Ventricles | 808.16 (150.14) | 788.25 (150.29)
Statistical Analysis 1: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Whole Brain: Analysis was based on RCRM using unstructured covariance matrix: MRI Whole Brain (Derived) = Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p = 0.25, RCRM; Difference in Annualized Rate of Change = 107.78, 95% CI 2-sided [-74.5 to 290.05], Standard Error of Mean 92.28
Statistical Analysis 2: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Bilateral Hippocampus: Analysis was based on RCRM using unstructured covariance matrix: MRI Bilateral Hippocampus = Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p = 0.58, RCRM; Difference in Annualized Rate of Change = 9.60, 95% CI 2-sided [-24.74 to 43.94], Standard Error of Mean 17.39
Statistical Analysis 3: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Ventricles: Analysis was based on RCRM using unstructured covariance matrix: MRI Ventricles = Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p = 0.93, RCRM; Difference in Annualized Rate of Change = 19.92, 95% CI 2-sided [-400.78 to 440.62], Standard Error of Mean 213.08

10. Secondary Outcome: Period A: Annualized Rate of Change in Tau-Based Cerebral Spinal Fluid (CSF) Biomarkers (Total Tau (tTau) and Phospho-tau (pTau)
Description: CSF biomarker tTau has been considered as a general marker of neurodegeneration. CSF phospho-tau is an indicator of neuronal injury and neurodegeneration. An elevation in levels of tau, as well as specific pTau species, is thought to be a marker for progressive cellular degeneration in AD. Annualized rate of change in tTau and pTau was estimated using RCRM.
Time Frame: Baseline up to approximately Week 416
Population: mITT population included all randomized participants who were mutation carriers and were treated with any amount of study drug. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Error); unit: picograms per milliliters (pg/mL)/year
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers
Number analyzed (Participants) | 48 | 42
picograms per milliliters (pg/mL)/year
  tTau | 4.91 (2.16) | 6.88 (2.19)
  pTau: number analyzed (Participants) | 44 | 40
  pTau | 0.84 (0.32) | 1.34 (0.33)
Statistical Analysis 1: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; tTau: Analysis was based on RCRM using unstructured covariance matrix: CSF tTau = Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p = 0.53, RCRM; Difference in Annualized Rate of Change = -1.97, 95% CI 2-sided [-8.17 to 4.23], Standard Error of Mean 3.09
Statistical Analysis 2: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; pTau: Analysis was based on RCRM using unstructured covariance matrix: CSF pTau = Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p = 0.28, RCRM; Difference in Annualized Rate of Change = -0.50, 95% CI 2-sided [-1.43 to 0.43], Standard Error of Mean 0.46

11. Secondary Outcome: Period A: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. An SAE is any AE that is fatal; life-threatening; requires or prolongs inpatient hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product(s); considered a significant medical event by the investigator. Pooled data has been reported for this outcome measure in order to maintain blinding of the participant's mutation status and treatment group.
Time Frame: From Baseline up to approximately Week 416
Population: Safety population included all randomized participants who received at least 1 dose of study drug; participants were grouped according to the actual treatment received and the mutation status.
Measure: Count of Participants; unit: Participants
Groups:
- Study Period A: Combined Blinded: All participants who were carriers and non-carriers of PSEN1 E280A mutation and who received either crenezumab, 720 mg, SC, Q2W, or 60 mg/kg, IV, Q4W, or crenezumab matching placebo for a minimum of 260 weeks during Period A are represented in this arm together for the purpose of maintaining blinding for participant's mutation status and treatment group.
Arm/Group | Study Period A: Combined Blinded
Number analyzed (Participants) | 251
Participants
  Participants with AEs | 251
  Participants with SAEs | 56

12. Secondary Outcome: Period A: Number of Participants Who Withdrew From the Study Treatment Due to AEs
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. Participants who withdrew from the study due to AEs are reported here. Pooled data has been reported for this outcome measure in order to maintain blinding of the participant's mutation status and treatment group.
Time Frame: From Baseline up to approximately Week 416
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period A: Combined Blinded
Number analyzed (Participants) | 251
Participants | 1

13. Secondary Outcome: Period A: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: AE=any unfavorable & unintended sign, symptom/disease temporally associated with use of an investigational product/other protocol-imposed intervention, regardless of attribution. Amyloid-related imaging abnormalities (ARIA)=spectrum of image abnormalities detected on MRI. Two types of ARIAs reported are: Amyloid-related Imaging Abnormalities-Edema/Effusion (ARIA-E)=MRI alterations thought to represent vasogenic edema (VE) & related extravasated fluid phenomena, & Amyloid-related Imaging Abnormalities-Hemosiderin Deposition (ARIA-H)=MRI alterations attributable to microhemorrhages (microbleeds [MBs]) & leptomeningeal hemosiderosis. Cerebral macrohemorrhages were read on MRI scans. Occurrence of pneumonia were verified by imaging (e.g., chest X-ray). Other AESIs were drug induced liver injury & suspected transmission of infectious agent via medicinal products. Pooled data has been reported for this outcome measure to maintain blinding of participant's mutation status & treatment group.
Time Frame: From Baseline up to approximately Week 416
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period A: Combined Blinded
Number analyzed (Participants) | 251
Participants
  ARIA-H | 6
  ARIA-E | 1
  Cerebral Macrohemorrhage | 0
  Drug Induced Liver Injury | 1
  Suspected Transmission of Infectious Agents via a Medicinal Product | 0
  Pneumonia | 0

14. Secondary Outcome: Period A: Number of Participants Injection Reactions and Infusion-related Reaction (IRRs)
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. Infusion and injection-related reactions were defined as any AEs that occurred during or within 24 hours after the study drug injection or infusion. Pooled data has been reported for this outcome measure in order to maintain blinding of the participant's mutation status and treatment group.
Time Frame: Baseline (Day 1) up to approximately Week 416
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period A: Combined Blinded
Number analyzed (Participants) | 251
Participants
  Injection Reaction | 92
  Infusion Related Reaction: number analyzed (Participants) | 200
  Infusion Related Reaction | 70

15. Secondary Outcome: Period A: Number of Participants With Anti-Crenezumab Antibodies
Description: The number of participants with positive results for ADA against crenezumab at any of the post-baseline assessment time-points were reported. Participants positive at any post-baseline time points were post-baseline evaluable participants determined to have "Treatment-induced ADAs" during the study period. Treatment-induced ADA = a participant with negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result.
Time Frame: Baseline up to approximately Week 260
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period A: Crenezumab - Mutation Carrier
Number analyzed (Participants) | 84
Participants | 5

16. Secondary Outcome: Period A: Cerebrospinal Fluid (CSF) Crenezumab Concentration
Time Frame: Predose: Baseline (Day 1), Weeks 104 and 260; early termination visit and unscheduled visit (up to approximately Week 416)
Population: PK-evaluable population included all safety-evaluable participants with at least 1 plasma sample, provided sufficient dosing information (dose and dosing time) is available. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliters (µg/ml)
Arm/Group | Study Period A: Crenezumab - Mutation Carrier
Number analyzed (Participants) | 36
micrograms per milliliters (µg/ml)
  Baseline (Day 1): number analyzed (Participants) | 25
  Baseline (Day 1) | NA (NA) — The data was not evaluable as the samples were below lower limit of quantification (BLLQ).
  Week 104 | 0.198 (81.6)
  Week 260: number analyzed (Participants) | 27
  Week 260 | 0.311 (214.6)
  Early Termination Visit: number analyzed (Participants) | 22
  Early Termination Visit | 0.238 (190.4)
  Unscheduled Visit: number analyzed (Participants) | 1
  Unscheduled Visit | 2.23 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable.

17. Secondary Outcome: Period A: Serum Crenezumab Concentration
Time Frame: Baseline (Day 1), Weeks 4, 12, 16, 17, 26, 38, 52, 78, 104, 128, 130, 156, 180, 182, 208, 232, 234, 260, 284, 312, 336, 364, 388, early termination visit and unscheduled visit (up to approximately Week 416)
Population: PK-evaluable population included all safety-evaluable participants with at least 1 plasma sample, provided sufficient dosing information (dose and dosing time) is available. Number analyzed is the number of participants with data available for analysis at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/ml
Arm/Group | Study Period A: Crenezumab - Mutation Carrier
Number analyzed (Participants) | 84
µg/ml
  Baseline (Day 1): number analyzed (Participants) | 80
  Baseline (Day 1) | NA (NA) — The data was not evaluable as the samples were BLLQ.
  Week 4 | 69.2 (39.1)
  Week 12 | 93.9 (51.8)
  Week 16: number analyzed (Participants) | 47
  Week 16 | 85.8 (37.2)
  Week 17: number analyzed (Participants) | 46
  Week 17 | 114 (37.3)
  Week 26: number analyzed (Participants) | 82
  Week 26 | 96.5 (86.3)
  Week 38: number analyzed (Participants) | 81
  Week 38 | 98.0 (121.6)
  Week 52: number analyzed (Participants) | 82
  Week 52 | 82.9 (285.3)
  Week 78: number analyzed (Participants) | 82
  Week 78 | 75.9 (777.0)
  Week 104: number analyzed (Participants) | 83
  Week 104 | 86.2 (680.2)
  Week 128: number analyzed (Participants) | 5
  Week 128 | 124 (28.6)
  Week 130: number analyzed (Participants) | 78
  Week 130 | 72.3 (1514.9)
  Week 156: number analyzed (Participants) | 82
  Week 156 | 80.7 (1445.4)
  Week 180: number analyzed (Participants) | 26
  Week 180 | 56.1 (3140.6)
  Week 182: number analyzed (Participants) | 55
  Week 182 | 85.5 (1135.4)
  Week 208: number analyzed (Participants) | 80
  Week 208 | 94.3 (983.0)
  Week 232: number analyzed (Participants) | 60
  Week 232 | 69.4 (3990.1)
  Week 234: number analyzed (Participants) | 21
  Week 234 | 62.3 (2724.2)
  Week 260: number analyzed (Participants) | 79
  Week 260 | 101 (1417.7)
  Week 284: number analyzed (Participants) | 66
  Week 284 | 131 (690.6)
  Week 312: number analyzed (Participants) | 53
  Week 312 | 116 (645.0)
  Week 336: number analyzed (Participants) | 30
  Week 336 | 117 (544.7)
  Week 364: number analyzed (Participants) | 16
  Week 364 | 227 (38.2)
  Week 388: number analyzed (Participants) | 11
  Week 388 | 162 (79.8)
  Early Termination Visit: number analyzed (Participants) | 77
  Early Termination Visit | 223 (135.5)
  Unscheduled: number analyzed (Participants) | 1
  Unscheduled | 98.4 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not evaluable.

18. Secondary Outcome: Period A: Annualized Rate of Change in Plasma Concentrations of Amyloid Beta 1(Aβ1)-40 and Amyloid Peptide Beta 42 (Aβ1-42)
Description: Amyloid beta is a peptide fragment of the amyloid precursor protein. The annualized rate of change in plasma concentration of Aβ1-40 and Aβ1-42 were estimated using a linear mixed effects model with random intercept and slope.
Time Frame: Baseline up to approximately Week 416
Population: as for outcome 2
Measure: Mean (Standard Error); unit: (pg/mL)/year
Arm/Group | Study Period A: Crenezumab - Mutation Carrier | Study Period A: Placebo - Mutation Carriers
Number analyzed (Participants) | 84 | 84
(pg/mL)/year
  Aβ1-40 | 6836.37 (236.49) | -686.18 (234.84)
  Aβ1-42 | 509.44 (17.74) | -46.59 (17.61)
Statistical Analysis 1: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Aβ1-40: Analysis was based on RCRM using unstructured covariance matrix: APlasma Amyloid Beta 1-40 =Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p < 0.0001, RCRM; Difference in Annualized Rate of Change = 7522.55, 95% CI 2-sided [6903.44 to 8141.65], Standard Error of Mean 313.17
Statistical Analysis 2: Comparison: Study Period A: Crenezumab - Mutation Carrier vs Study Period A: Placebo - Mutation Carriers; Aβ1-42: Analysis was based on RCRM using unstructured covariance matrix: Plasma Amyloid Peptid Beta 42 =Treatment * Analysis Year + IxRS defined Age Group + IxRS defined Education History + IxRS defined APOE4 Carrier Status + IxRS defined CDR Global Score; Test type: Superiority; p < 0.0001, RCRM; Difference in Annualized Rate of Change = 556.03, 95% CI 2-sided [508.63 to 603.44], Standard Error of Mean 23.98

19. Secondary Outcome: Period B: Number of Participants With AEs and SAEs
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. An SAE is any AE that is fatal; life-threatening; requires or prolongs inpatient hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product(s); considered a significant medical event by the investigator. During Study Period B, after the results of Study Period A were available, participants had an option to learn their mutation carrier status. Since all participants did not choose to learn their mutation status, pooled data has been presented for this outcome measure in order to maintain blinding of the participant's mutation status and treatment group assigned.
Time Frame: From Day 1 (Period B) up to 67 weeks
Population: Safety population included all randomized participants who received at least 1 dose of study drug in Study Period B; participants are grouped according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Study Period B: Combined Blinded: All participants who were carriers and non-carriers of PSEN1 E280A mutation and who received either crenezumab 720 mg, SC, Q2W, or 60 mg/kg, IV, Q4W, or crenezumab matching placebo for up to 51 weeks during Period B are represented in this arm together for the purpose of maintaining blinding for participant's mutation status and treatment group.
Arm/Group | Study Period B: Combined Blinded
Number analyzed (Participants) | 219
Participants
  Participants with AEs | 219
  Participants with SAEs | 12

20. Secondary Outcome: Period B: Number of Participants Who Withdraw From the Study Treatment Due to AEs
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. During Study Period B, after the results of Study Period A were available, participants had an option to learn their mutation carrier status. Since all participants did not choose to learn their mutation status, pooled data has been presented for this outcome measure in order to maintain blinding of the participant's mutation status and treatment group assigned.
Time Frame: From Day 1 (Period B) up to 67 weeks
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period B: Combined Blinded
Number analyzed (Participants) | 219
Participants | 0

21. Secondary Outcome: Period B: Number of Participants With AESIs: ARIA-E, ARIA-H, Cerebral Macrohemorrhages, and Pneumonia
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. ARIA are a spectrum of image abnormalities detected on MRI. The two types of ARIA reported will include: ARIA-E: refers to the MRI alterations thought to represent VE and related extravasated fluid phenomena, and ARIA-H: refers to the MRI alterations attributable to MBs and leptomeningeal hemosiderosis. Cerebral macrohemorrhages will be read on MRI scans. Occurrence of pneumonia will be verified by imaging (e.g., chest X-ray). During Study Period B, after the results of Study Period A were available, participants had an option to learn their mutation carrier status. Since all participants did not choose to learn their mutation status, pooled data has been presented for this outcome measure in order to maintain blinding of the participant's mutation status and treatment group assigned.
Time Frame: From Day 1 (Period B) up to 67 weeks
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period B: Combined Blinded
Number analyzed (Participants) | 219
Participants
  Pneumonia | 1
  ARIA-H | 0
  ARIA-E | 0
  Cerebral Macrohemorrhage | 0
  Drug Induced Liver Injury | 0
  Suspected Transmission of Infectious Agents via a Medicinal Product | 0

22. Secondary Outcome: Period B: Number of Participants With Injection Reactions and IRRs
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. Infusion and injection-related reactions are defined as any AEs that occurred during or within 24 hours after the study drug injection or infusion. During Study Period B, after the results of Study Period A were available, participants had an option to learn their mutation carrier status. Since all participants did not choose to learn their mutation status, pooled data has been presented for this outcome measure in order to maintain blinding of the participant's mutation status and treatment group assigned.
Time Frame: From Day 1 (Period B) up to 67 weeks
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period B: Combined Blinded
Number analyzed (Participants) | 219
Participants
  Injection Reaction | 1
  Infusion Related Reaction | 12

ADVERSE EVENTS:
Time Frame: Period A: Baseline up to approximately 416 weeks; Period B: Day 1 (Period B) up to 67 weeks. To protect the mutation status in Periods A & B, for deaths & SAEs: data are reported in each arm under system organ class (SOC) of General Disorders & participant level data are reported in Combined Blinded arms only. All arms were considered to be at Risk for all deaths/SAEs although participant level data are reported in Combined blinded arms only. Data for OAEs are reported under SOC's for all arms.
Description: Safety population used for Period A&B. Period A= 1 participant excluded from safety population for not meeting 1 of the eligibility criteria prior to treatment start.
  During Period B, after Period A results were available, participants had an option to learn their mutation status. All participants did not choose to learn their mutation status. Hence, pooled data has been presented to maintain blinding of participant's mutation status & treatment assignment. OAEs=Other Adverse Events.
Groups:
- Study Period A: Crenezumab - Mutation Carriers: Participants with PSEN1 E280A mutation, received crenezumab, 720 mg, SC, Q2W, or 60 mg/kg, IV, Q4W, for a minimum of 260 weeks during Period A.
- Study Period A: Placebo - Mutation Carriers: Participants who were PSEN1 E280A mutation carriers, received crenezumab matching placebo SC, Q2W, or IV, Q4W, for a minimum of 260 weeks during Period A.
- Study Period A: Combined Blinded: All participants who were carriers and non-carriers of PSEN1 E280A mutation and who received either crenezumab placebo 720 mg, SC, Q2W, or 60 mg/kg, IV, Q4W, or crenezumab matching for a minimum of 260 weeks during Period A are represented in this arm together for the purpose of maintaining blinding for participant's mutation status and treatment group.
- Study Period B: Placebo: Participants who were non-carriers of PSEN1 E280A mutation and who received crenezumab matching placebo in Period A were given an option to continue receiving crenezumab matching placebo SC, Q2W or IV, Q4W in Study Period B, for up to 51 weeks.
Arm/Group | Study Period A: Crenezumab - Mutation Carriers | Study Period A: Placebo - Mutation Carriers | Study Period A: Placebo - Non-Carriers of Mutation | Study Period A: Combined Blinded | Study Period B: Crenezumab | Study Period B: Placebo | Study Period B: Combined Blinded
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/84 | 0/83 | 0/251 | 0/147 | 0/72 | 1/219
Serious Adverse Events (participants affected / at risk) | 23/84 | 21/84 | 12/83 | 56/251 | 9/147 | 3/72 | 12/219
Other Adverse Events (participants affected / at risk) | 84/84 | 84/84 | 83/83 | 251/251 | 95/147 | 54/72 | 149/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Period A: Crenezumab - Mutation Carriers (N=84) | Study Period A: Placebo - Mutation Carriers (N=84) | Study Period A: Placebo - Non-Carriers of Mutation (N=83) | Study Period A: Combined Blinded (N=251) | Study Period B: Crenezumab (N=147) | Study Period B: Placebo (N=72) | Study Period B: Combined Blinded (N=219)
Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 12 (13) | 0 (0) | 0 (0) | 5 (5)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 2 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Nervous system disorders (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (2)
Social circumstances (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
General disorders and administration site conditions (General disorders) | 23 (30) | 21 (22) | 12 (14) | 2 (2) | 9 (18) | 3 (5) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Study Period A: Crenezumab - Mutation Carriers (N=84) | Study Period A: Placebo - Mutation Carriers (N=84) | Study Period A: Placebo - Non-Carriers of Mutation (N=83) | Study Period A: Combined Blinded (N=251) | Study Period B: Crenezumab (N=147) | Study Period B: Placebo (N=72) | Study Period B: Combined Blinded (N=219)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 14 (25) | 9 (12) | 8 (13) | 31 (50) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders (Cardiac disorders) | 8 (12) | 11 (13) | 6 (8) | 25 (33) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 15 (18) | 10 (21) | 20 (25) | 45 (64) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders (Endocrine disorders) | 5 (5) | 8 (8) | 5 (5) | 18 (18) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 55 (141) | 60 (152) | 54 (144) | 166 (437) | 20 (25) | 11 (11) | 31 (36)
General disorders and administration site conditions (General disorders) | 39 (82) | 39 (100) | 43 (91) | 121 (273) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations (Infections and infestations) | 84 (772) | 81 (839) | 83 (854) | 248 (2465) | 46 (66) | 29 (44) | 75 (110)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 60 (185) | 58 (190) | 54 (161) | 174 (536) | 23 (33) | 10 (11) | 33/129 (44)
Investigations (Investigations) | 17 (21) | 15 (20) | 17 (33) | 49 (74) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 35 (57) | 22 (31) | 32 (47) | 89 (135) | 8 (9) | 6 (6) | 14 (15)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 64 (177) | 65 (220) | 66 (284) | 195 (681) | 17 (19) | 19 (23) | 36 (42)
Nervous system disorders (Nervous system disorders) | 66 (297) | 70 (311) | 62 (309) | 198 (917) | 27 (45) | 14 (18) | 41 (63)
Psychiatric disorders (Psychiatric disorders) | 43 (109) | 44 (111) | 44 (105) | 131 (325) | 21 (27) | 4 (5) | 25 (32)
Renal and urinary disorders (Renal and urinary disorders) | 18 (28) | 15 (21) | 12 (15) | 45 (64) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 24 (56) | 35 (82) | 39 (100) | 98 (238) | 20 (23) | 10 (11) | 30 (34)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 15 (20) | 17 (23) | 22 (24) | 54 (67) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 38 (91) | 41 (75) | 48 (93) | 127 (259) | 8 (10) | 7 (7) | 15 (17)
Vascular disorders (Vascular disorders) | 15 (17) | 20 (26) | 18 (23) | 53 (66) | 0 (0) | 0 (0) | 0 (0)
Eye disorders (Eye disorders) | 20 (25) | 10 (17) | 14 (17) | 44 (59) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 11 (11) | 12 (13) | 28 (30) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT01998841/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT01998841/SAP_001.pdf